CLINICAL TRIAL: NCT01994317
Title: Use of an Algorithm to Determine IV Sedation Dosing During First-trimester Surgical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFPRF7-6
Record Dates: First submitted 2013-11-01; First posted 2013-11-25 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Pregnancy, Unplanned
MeSH Terms: interventions — Algorithms; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard sedation dose (Active Comparator): IV sedation dose calculated using current standard of care
  Interventions: Other: Standard care
- Algorithm (Experimental): IV sedation dose calculated by study algorithm
  Interventions: Other: Algorithm

INTERVENTIONS:
Other: Algorithm — IV sedation dosing calculated by algorithm
  Arms: Algorithm
Other: Standard care — IV sedation dosing calculated by standard care.
  Arms: Standard sedation dose

SUMMARY:
This study aims to compare an algorithm for IV sedation dosing to the current standard of care in patients undergoing first trimester surgical abortion. The primary outcome is subjects' pain score with suction curettage on a 0-100 21-point scale. Secondary outcomes include pain scores with cervical dilation and 15 minutes post-procedure, subjective pain ratings, incidents of side effects and adverse events, the frequency of additional doses of medication, recovery room time, and physician assessment of and satisfaction with pain control. Investigators hypothesize that this algorithm will result in improved pain control, decreased frequency of additional medication doses, improved patient and physician satisfaction, without differences in side effects, adverse events or recovery room time.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older seeking surgical abortion at Planned Parenthood League of Massachusetts (PPLM)
* Gestational age less than or equal to 13+6, confirmed by ultrasound
* Eligible for surgical abortion according to PPLM protocols
* Eligible for IV sedation per PPLM protocol, and desiring IV sedation for pain management

Exclusion Criteria:

* Choice of local anesthesia for pain control
* Hypersensitivity to midazolam or fentanyl
* Ineligible for IV sedation per PPLM protocol
* Need for cervical ripening with either misoprostol or mechanical priming agent (laminaria/Dilapan)
* Unable or unwilling to complete required study procedures
* Previous participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain with suction curettage | Measured on Day 1 (day of enrollment), immediately (within one minute) after completion of suction curettage and speculum removal
  Subjects' pain score with suction curettage on a 0-100 21-point scale

SECONDARY OUTCOMES:
Pain with paracervical block | Measured on Day 1 (day of enrollment), immediately after paracervical block
  Pain with paracervical block will be measured (a) on a 21-point 0 to 100 scale (in increments of five), and (b) on a subjective scale of "no pain, mild pain, moderate pain or severe pain." Pain will be measured immediately after paracervical block.
Pain with cervical dilation | Measured on Day 1 (day of enrollment), immediately after cervical dilation
  Pain with cervical dilation will be measured (a) on a 21-point 0 to 100 scale (in increments of five), and (b) on a subjective scale of "no pain, mild pain, moderate pain or severe pain." Pain with cervical dilation will be measured immediately after cervical dilation.
Post-operative pain | Measured on Day 1 (day of enrollment), 15 minutes post-operatively
  Post-operative pain will be measured (a) on a 21-point 0 to 100 scale (in increments of five), and (b) on a subjective scale of "no pain, mild pain, moderate pain or severe pain." Pain will be measured 15 minutes post-operatively when the patient is in the recovery room.
Patient satisfaction with pain control | Measured on Day 1 (day of enrollment), 15 minutes post-operatively
  Patients will be asked about their general satisfaction with pain control, what their pain was compared to what they expected, whether they would chose the same pain management strategy again, and whether they would recommend their strategy of pain management to a friend.
Side effects | Measured on Day 1 (day of enrollment), 15 minutes post-operatively
  Investigators will assess side effects for all patients, including nausea, vomiting, dizziness, and drowsiness.

OTHER OUTCOMES:
Doses given over the duration of the study | Measured on Day 1 (day of enrollment), intraoperatively
  To assess whether use of the algorithm changes physician's behavior in the standard care arm, investigators will also examine doses given over the duration of the study, to see if a "learning curve" develops among the physicians based on their experience with the algorithm.
Physician assessment of pain control | Measured on Day 1 (day of enrollment), post-operatively
  Investigators will also have the physician assess patients' pain control, whether they felt the dose was appropriate and how easy or difficult it was to determine the patients' doses of pain medication.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — PPLM
Locations (1):
- Planned Parenthood, Boston, Massachusetts, United States